CLINICAL TRIAL: NCT04264949
Title: E-lombactifs: Evaluation of the Impact a Smartphone Application on Adherence an Exercise Program in Chronic Low Back Pain
Acronym: E-lombactifs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RBHP 2019 LECHAUVE; 2019-A02191-56 (Other: 2019-A02191-56)
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic Low Back Pain; Physical activity; Adherence
MeSH Terms: conditions — Motor Activity | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group application (GA) (Experimental): benefit from conventional care in a rehabilitation center, therapeutic education program and education in the use of the smartphone application "mon coach dos"
  Interventions: Other: Education in the use of smartphone app (Mon coach dos); Other: conventional care
- Groupe conventional care (GCC) (Active Comparator): benefit from conventional care in a rehabilitation center and therapeutic education program
  Interventions: Other: conventional care

INTERVENTIONS:
Other: Education in the use of smartphone app (Mon coach dos) — In addition to conventional care and the therapeutic education program, GA will benefit from three education sessions (one per week) on the use of the smartphone app mon coach dos
  Arms: group application (GA)
Other: conventional care — conventional care and the therapeutic education program

SUMMARY:
The main objective is to assess the impact of smartphone application on adherence to a physical exercise program in chronic low back pain patients.

Adherence to a physical exercise program will be assessed at the start of the protocol, at three weeks and six months.

A control group will benefit from conventional care in a rehabilitation center and an intervention group will benefit from a conventional care in a rehabilitation center accompanied by education in the use of a smartphone application including physical exercises and information about low back pain.

The hypothesis of the search is that adherence is better in intervention group than control group at 6 months due to education in the use of smartphone application.

ELIGIBILITY:
Inclusion Criteria:

* Adult People
* With nonspecific chronic low back pain (according to the definition of the HAS)
* Covered under the national health insurance
* Giving informed written consent to participate in the study

Exclusion Criteria:

* Patient who do not meet the diagnostic criteria according to the definition of HAS
* Behavioral disorders or comprehension difficulties making assessment impossible
* Patient with a contraindication to physical exercise for medical reasons
* Patient under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
EARS : exercise adherence rating scale | day1
  EARS assess the adherence in physical activity program.
EARS : exercise adherence rating scale | day 15
  EARS assess the adherence in physical activity program.
EARS : exercise adherence rating scale | day 180
  EARS assess the adherence in physical activity program.

SECONDARY OUTCOMES:
OSWESTRY questionnaire | day1, day 15, day 180
  Disability is measured by OSWESTRY
EPAP questionnaire | day1, day 15, day 180
  The perceived barriers to and facilitators of physical activity are measured by EPAP
Pain measurment: numeric scale | day1, day 15, day 180
  The pain is measured by numeric scale
6 minutes' walk test (6MWT) | day1, day 15, day 180
  Aerobic and functional capacities are measured by 6 minutes' walk test (6MWT)
aerobic capacities | day1, day 15, day 180
  aerobic capacities are measured by sub maximal ergocycle test
muscular endurance | day1, day 15, day 180
  the muscular endurance of the erector muscles of the spine is measured by Sorensen test
muscular endurance of the flexor muscles of the spine | day1, day 15, day 180
  the muscular endurance of the flexor muscles of the spine is measured by ITO test
muscular endurance of the extensor of the knee | day1, day 15, day 180
  the muscular endurance of the extensor of the knee is measured by Killy test
Core measurment | day1, day 15, day 180
  Core is measured by plank test
Flexibility on posterior chain | day1, day 15, day 180
  Flexibility on posterior chain is measured by DDS test
Mobility on posterior chain | day1, day 15, day 180
  Mobility on posterior chain is measured by Schober test

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Lechauve, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Lechauve JB, Dobija L, Pereira B, Grolier M, Goldstein A, Lanhers C, Coudeyre E. Evaluation of the impact of a smartphone application on adherence to home exercise program for people with chronic low back pain: research protocol for a pilot randomised controlled trial. BMJ Open. 2023 Mar 24;13(3):e062290. doi: 10.1136/bmjopen-2022-062290. PMID 36963800